CLINICAL TRIAL: NCT06869343
Title: A Randomized Controlled Trial of Early Versus Delayed Rehabilitation After Reverse Total Shoulder Arthroplasty for Proximal Humerus Fracture
Brief Title: Early Versus Delayed Rehabilitation After Reverse Total Shoulder Arthroplasty for Proximal Humerus Fracture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Foundation of Orthopedic Trauma (Other)
Responsible Party: Principal Investigator, Seth Yarboro, MD, Associate Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSR301914; FOT Grant ID 9024-2 (Other Grant/Funding Number: Foundation for Orthopaedic Trauma)
Record Dates: First submitted 2025-02-28; First posted 2025-03-11 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-03

CONDITIONS: Orthopedic Disorder; Humerus Fracture; Shoulder Arthroplasty; Reverse Shoulder Replacement
MeSH Terms: conditions — Musculoskeletal Diseases; Humeral Fractures | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Onset Physical Therapy (Active Comparator): Patients in this arm will begin post operative physical therapy at 2 weeks after procedure.
  Interventions: Other: Physical Therapy
- Delayed Onset Physical Therapy (Active Comparator): Patients in this arm will begin post operative physical therapy at 6 weeks after procedure.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — Subjects will begin physical therapy at either 2 or 6 weeks s/p a rTSA.

SUMMARY:
Proximal humerus fractures can be a debilitating injury in the elderly, impacting the ability to function independently or complete activities of daily living due to pain and restricted shoulder motion. Evidence has shown that reverse total shoulder arthroplasty (rTSA) is an effective option to improve pain and function for patients with acute displaced proximal humerus fractures. Given that patients undergoing rTSA for proximal humerus fractures typically experience worse functional outcomes, worse patient-reported outcomes, and higher rates of complication compared to those with elective indications for surgical intervention, it is critical to determine a secure path to recovery for these patients after surgery. Early rehabilitation has been proposed to be safe and effective for patients who undergo rTSA for elective indications; however, there is a paucity of research evaluating safety and effectiveness of timing of rehabilitation for rTSA patients in the trauma setting. Currently, there exists a great variability in postoperative rehabilitation protocols across orthopaedic practices. This study's objective is to determine the safety and effectiveness of early postoperative rehabilitation on the outcomes and postoperative complications of patients undergoing rTSA for proximal humerus fractures in order to provide more specific recommendations for this patient population.

DETAILED DESCRIPTION:
The overarching goal is to better understand the impact of timing of initiation of rehabilitation on functional and patient reported outcomes on patients undergoing rTSA in the trauma setting.

Specifically, the investigators will conduct a pilot study in the form of a randomized controlled trial to evaluate whether, in patients undergoing rTSA for proximal humerus fracture, early rehabilitation yields a significant difference in range of motion, patient-reported outcomes, or postoperative complications compared to those who undergo delayed rehabilitation. The specific aims are:

Aim 1: To compare the range of motion and patient reported outcomes between early and delayed rehabilitation in patients undergoing rTSA for proximal humerus fracture by conducting a randomized trial. The investigators will enroll patients in a randomized controlled trial postoperatively that will allocate patients to begin physical rehabilitation early (two weeks after operation) or delayed (six weeks after operation). In-person clinic visits and radiographs will occur at multiple time points (six weeks, three months, and six months) postoperatively. The investigators hypothesize that patients undergoing rTSA for proximal humerus fracture participating in early rehabilitation will have no difference in range of motion (forward flexion, abduction) or patient reported outcomes American Shoulder Elbow Surgeons Shoulder Score Constant score.

Aim 2: To compare the rates of postoperative complications between early and delayed rehabilitation in patients undergoing rTSA for proximal humerus fracture. Investigators will conduct chart reviews as well as in-person clinic visits and radiographs at multiple time points postoperatively. Investigators hypothesize that there will be no difference in rates of postoperative complications between early and delayed rehabilitation groups.

The expected outcome of this study is an enhanced understanding of the impact of rehabilitation after proximal humerus fracture, and the degree to which timing of initiation of therapy impacts patient outcomes. This will have a positive impact because it creates a foundation for developing rehabilitation protocols in this population.

ELIGIBILITY:
Inclusion Criteria:

* aged 50-85 undergo reverse Total Shoulder Arthroplasty by a single surgeon for proximal humerus fractures

Exclusion Criteria:

* previous rTSA to ipsilateral shoulder
* undergoing elective rTSA
* Prisoners
* unwilling to be randomized
* unwilling or unable to attend follow up visits

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of Range of motion of shoulder Forward Flexion using a goniometer | 2 week, 6 week, 3 month, and 6 month
  A goniometer will be used to measure forward flexion of the shoulder.

CONTACTS AND LOCATIONS:
Overall Officials: Seth Yarboro, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Medical Center, Charlottesville, Virginia, United States